CLINICAL TRIAL: NCT00848237
Title: HALO Patient Registry: Ablation of Barrett's Esophagus, A Multi-Center Patient Registry
Brief Title: HALO Patient Registry: Ablation of Barrett's Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-500
Record Dates: First submitted 2007-12-20; First posted 2009-02-20 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Barrett Esophagus
Keywords: Barrett's Esophagus; Dysplasia; Intestinal Metaplasia
MeSH Terms: conditions — Barrett Esophagus | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): All Patients with Barrett's esophagus or Intestinal metaplasia which is visible endoscopically or histologically may be treated with the Radiofrequency ablation system.
  Interventions: Device: Radiofrequency Ablation (HALO Ablation Systems)

INTERVENTIONS:
Device: Radiofrequency Ablation (HALO Ablation Systems) — Subjects undergo ablation procedures (circumferential or focal) plus standard anti-secretory drug therapy (proton pump inhibitor, PPI). All Patients undergo endoscopy with biopsy in a Physician prescribed surveillance pattern after a negative biopsy.
  Other Names: HALO 90; HALO 360

SUMMARY:
The HALO Patient Registry is a prospective/retrospective, multi-center patient registry. It provides a framework for treatment and follow-up of patients with Barrett's esophagus (non-dysplastic IM, LGD and HGD). The primary objective is to provide a tool for participating physician investigators to collect outcomes data related to the use of the HALO Ablation Systems.

DETAILED DESCRIPTION:
Summary The HALO Patient Registry provides a framework for treatment and follow-up of patients with Barrett's esophagus (non-dysplastic IM, LGD and HGD). The primary objective is to provide a tool for participating physician investigators to collect outcomes data related to the use of the HALO Ablation Systems.

Protocol Design:

This is a prospective, multi-center patient Registry. Sites may choose to also retrospectively enroll previously treated patients (after obtaining informed consent) and enter retrospective data into case report forms on-line. "Retrospective data collection" is defined as any data other than patient history collected prior to signing of the informed consent. A set of case report forms (CRFs) is provided along with this protocol to track outcomes. The CRFs may be completed and retained on site, but the site is recommended to utilize the internet-based data entry system.

ELIGIBILITY:
Inclusion Criteria:

* Must be a candidate for ablation of Barrett's esophagus with the HALO Ablation System.
* Must agree to the proposed follow-up schedule and provide informed consent for participation.

Exclusion Criteria:

* Pregnancy
* Prior radiation therapy to the esophagus
* Esophageal varices at risk for bleeding
* Prior Heller Myotomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5521 (Actual)
Dates: Start 2007-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Shaheen, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Gastrointestinal Associates and sites across the US, Knoxville and Other US Cities, California, United States

REFERENCES:
- [Result] Shaheen NJ, Kim HP, Bulsiewicz WJ, Lyday WD, Triadafilopoulos G, Wolfsen HC, Komanduri S, Chmielewski GW, Ertan A, Corbett FS, Camara DS, Rothstein RI, Overholt BF. Prior fundoplication does not improve safety or efficacy outcomes of radiofrequency ablation: results from the U.S. RFA Registry. J Gastrointest Surg. 2013 Jan;17(1):21-8; discussion p.28-9. doi: 10.1007/s11605-012-2001-8. Epub 2012 Sep 11. PMID 22965650

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 5521
Completed | 4982
Not Completed | 539

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 5521
Age, Categorical [Number; unit: participants] — Note: 6 subjects: Age unknown
  participants
    <=18 years | 1
    Between 18 and 65 years | 3235
    >=65 years | 2279
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1469
  Male | 4052
Region of Enrollment [Number; unit: participants]
  United States | 5521

OUTCOME MEASURES:

1. Primary Outcome: Endoscopic Clearance Rate for Barrett's Esophagus-Percentage of Patients With no Endoscopically Visible Barrett's Esophagus at 1 Year Follow-up
Description: % of patients with 100 % resolution at 1 year follow-up. This endpoint is a visual and not reliable or accurate. A better measure of clearance of Barrett's esophagus is based on biopsies.
Time Frame: 1 year
Population: 4011 subjects provided the answers
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 4011
percentage of participants | 62.1

2. Primary Outcome: Histological Clearance Rate for Intestinal Metaplasia (CE-IM)
Description: Percentage of patients with no histological evidence of intestinal metaplasia at 1 year follow-up
Time Frame: 1 year
Population: 4118 provided biopsies at least 1 year post RFA
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 4118
percentage of participants | 85.5

3. Primary Outcome: Histological Clearance Rate for Dysplasia (CE-D)
Description: percentage of patients with baseline dysplasia who have no histological evidence of dysplasia at 1 year follow-up
Time Frame: 1 year
Population: 4118 provided biopsies at least 1 year post RFA and non dysplasia subjects from 4118 were removed for CE-D analysis
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 2224
percentage of participants | 93.5

4. Primary Outcome: Percentage of Patients With Sub-squamous Intestinal Metaplasia at 1 Year Follow up
Description: Percentage of patients at 1 year follow-up with sub-squamous intestinal metaplasia, with or without dysplasia, that is covered completely by an intact layer of squamous epithelium with no communication with the surface
Time Frame: 1 year
Measure: Number; unit: percentage of patients with SSIM
Arm/Group | Treatment
Number analyzed (Participants) | 5521
percentage of patients with SSIM | 2.7

5. Primary Outcome: Patient Quality of Life Questionnaire Results: Change From Baseline to 12 Month
Description: Patient who completed both baseline and follow-up Quality of Life: Scores (0-10) of quality of life at baseline and 12 month follow-up were measured and changes were calculated ( 12 months minus baseline) in: concerns about the condition of esophagus, negative impact on life and esophageal cancer worry. Scale range is 0-10, 0 is min and 10 is max. Higher value represent worse outcome (such as higher concern about the condition of esophagus, negative impact on life and higher esophageal cancer worry).
Time Frame: 12 month
Population: 943 subjects completed both baseline and follow up quality of life life survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 943
units on a scale
  Changes:concern about the condition of esophagus | -2.7 (3.2)
  Negative impact on life | -1.9 (3.0)
  Esophageal cancer worry | -2.8 (3.4)

6. Primary Outcome: Adverse Event Incidence
Description: Adverse and Serious Adverse event with Definite device relationship
Time Frame: 12 month
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 5521
participants | 66

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 24/5521
Other Adverse Events (participants affected / at risk) | 42/5521
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=5521)
Pain, Nausea, vomitting, fullness, abdominal discomfort (Injury, poisoning and procedural complications) | 6
Dysphagia and/or Odynophagia (Injury, poisoning and procedural complications) | 2
aspiration (Injury, poisoning and procedural complications) | 1
Dysphagia/Upper GI Bleed (Injury, poisoning and procedural complications) | 1
Esophageal spasms (Injury, poisoning and procedural complications) | 1
Esophagitis and/or Ulceration (Injury, poisoning and procedural complications) | 2
Fever (Injury, poisoning and procedural complications) | 2
Hematemesis (Injury, poisoning and procedural complications) | 1
Melena (Injury, poisoning and procedural complications) | 3
Mucosal Tear / Laceration (Injury, poisoning and procedural complications) | 1
Perforation (Injury, poisoning and procedural complications) | 1
Stricture and/or dysphagia requiring dilatation (Injury, poisoning and procedural complications) | 2
Upper GI Bleeding (Injury, poisoning and procedural complications) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=5521)
Catheter interaction with existing sutures (Injury, poisoning and procedural complications) | 1
Dysphagia and/or Odynophagia (Injury, poisoning and procedural complications) | 4
Esophageal spasms (Injury, poisoning and procedural complications) | 1
Esophagitis and/or Ulceration (Injury, poisoning and procedural complications) | 4
Hematemesis (Injury, poisoning and procedural complications) | 1
Mallory-weiss tear (Injury, poisoning and procedural complications) | 1
Mucosal Tear / Laceration (Injury, poisoning and procedural complications) | 14
Mucosal trauma (Injury, poisoning and procedural complications) | 1
Oxygen desaturation (Injury, poisoning and procedural complications) | 1
Pain, Nausea, vomitting, fullness, abdominal discomfort (Injury, poisoning and procedural complications) | 12
Prior Stricture worsen by RFA (Injury, poisoning and procedural complications) | 1
Sizing Balloon did not work (Injury, poisoning and procedural complications) | 1
Stricture - no dilatation (Injury, poisoning and procedural complications) | 12
Stricture and/or dysphagia requiring dilatation (Injury, poisoning and procedural complications) | 37
Stricture requiring dilatation- History EMR or Stricture (Injury, poisoning and procedural complications) | 2
Upper GI Bleeding (Injury, poisoning and procedural complications) | 5

LIMITATIONS AND CAVEATS:
Endoscopic clearance rate for Barrett's esophagus-Percentage of patients with no endoscopically visible Barrett's esophagus at 1 year follow-up: This endpoint is a visual and not reliable or accurate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less